CLINICAL TRIAL: NCT02865291
Title: Safety and Effectiveness Evaluation of the ForConti Fecal Management System - Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: ForConti Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CD-14-001
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ForConti device (Experimental): Use the device up to 12 hours/day for 4 weeks
  Interventions: Device: ForConti device

INTERVENTIONS:
Device: ForConti device

SUMMARY:
The ForConti Fecal Incontinence Management System (FIMS) is indicated for the management of accidental bowel leakage due to bowel incontinence. The ForConti FIMS is designed for self-insertion to seal and help prevent the involuntary leakage of stool, liquids and gases from the rectum.

The purpose of the study is to demonstrate that the ForConti FIMS is safe and that it improves management of fecal incontinence and improves quality of life.

Patients will record bowel events in a daily diary over a 6 week period, which includes 2 weeks without using the device followed by 4 weeks using the device. Quality of Life questionnaire will be completed before and after use of the device. Stool leakage data collected when the device is not being used will be compared with data collected during use of the device to determine effectiveness.

DETAILED DESCRIPTION:
There are several devices for treating bowel incontinence. However, available devices have limited success. Sphincter bulking agents and electrical stimulation did not demonstrate effectiveness in clinical studies. Anal plugs did show some effectiveness but are associated with discomfort and pain. Hence, patients prefer not to use them.

The main reason for pain and discomfort with the current available anal plugs is the plug location within the anus below the dentate line. This part of the anus which is highly sensitive it causes discomfort and pain to the user. The advantage of the ForConti device is that it is designed to be located at a more inner section of the anal canal, above the dentate line, which is much less sensitive thus does not cause discomfort to the user.

This is a prospective, feasibility, non-randomized, single-arm, self-controlled study for preliminary safety and effectiveness. Total duration of the study for each patient will be 8 weeks, including follow-up.

The study will be conducted on up to 20 patients suffering from accidental bowel leakage due to bowel incontinence and who meet all of the inclusion criteria and none of the exclusion criteria. Following first 5 cases, interim preliminary safety analysis was conducted and a report submitted to Ministry of Health for approval to continue the study. Approval was granted.

Primary Safety: No device related serious adverse events. Secondary Safety: Minimal rate of device or procedure related adverse events (intra and post-operative complications) in the treatment or in the follow-up periods.

Effectiveness:

Demonstrate the effectiveness of the system by:

A Relative Percentage Change in Episodes of Accidental Bowel Leakage (ABL, FI episodes) Determined by Comparing Active Weeks to Control Weeks Results as measured by Daily Diary Recordings.

Active Weeks are the 3rd and 4th week of study treatment period and the Control Weeks are the baseline 2 weeks assessment period before starting treatment.

Other Measurements:

Usability: Evaluation of SUS Scores Quality of Life: Recording and Evaluation of a validated symptom-specific Fecal Incontinence Quality of Life (FIQoL) Questionnaire Number of incontinence days while using the device during the two-week assessment period, as compared to the baseline two-week assessment period.

The ForConti FIMS includes 2 main parts: the inserted part and the insertion system. The inserted part includes a balloon and a pulling string and the insertion system includes the applicator, plunger and the inflator. The balloon is a flexible biocompatible, silicone-based, oval-shaped, furled component. It is designed to be located in the rectum by an applicator and to be filled with a pre-determined amount of air to gain its final shape. The silicone surface is equipped with silicone gags which provide better sustainability in the rectum.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the informed consent form and is willing to participate in the clinical study and data collection. Patient has the ability to self-manage insertion and removal of the device.
2. Patient age is between 18 and 85 years old
3. History of fecal incontinence for at least 6 months
4. A minimum of four incontinence episodes during the 2-week baseline period
5. Patient colon surveillance must be in compliance with the Ministry of Health National Program American Cancer Society colon for the Early Detection of Colorectal Cancer screening guidelines.
6. Patient comprehends study meaning & is capable of carrying out study duties.

Exclusion Criteria:

1. Spinal cord injury or other major neurological diagnosis
2. Known life threatening disease such as cancer, immune deficiency state
3. Significant cardiac arrhythmia
4. Pregnant or Breastfeeding
5. Inflammatory bowel disease
6. Anti-coagulants and anti-platelets treatment, except Aspirin (low dose: 75-100 mg/day)
7. Anorectal diseases: perianal abscess, active fistula, fissure, hemorrhoids grade 3 or 4, Pruritus ani or rectal bleeding
8. Chronic pelvic pain
9. Rectal surgery in past 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 6 weeks
  4 weeks of use and 2 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mark Beer-Gabel, MD — Sheba Medical Center; Josef Lysi, MD — Shaheed Ziaur Rahman Medical College

IPD SHARING:
Plan to Share IPD: No